CLINICAL TRIAL: NCT06464627
Title: Physical Activity Reduces Anxiety and Depression in Youth Affected by Displacement: a Randomized Controlled Trial of the Game Connect Program in Uganda
Acronym: Game Connect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Makerere University (Other); The University of New South Wales (Other); AVSI (Unknown); Olympic Refuge Foundation (Unknown)
Responsible Party: Principal Investigator, Davy Vancampfort, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10.05.2024
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity (Experimental): The project lasts 16 weeks and focuses on: improving skills and capacities of refugee and host community youth to support their psychosocial wellbeing and mental health through improved access to safe sport; developing a new/strengthened social and support network through safe sport, including those from diverse backgrounds among refugee and host community youth; working with and ensuring District Level officials appreciate and advocate for Sport for Protection activities.
  Interventions: Behavioral: Physical activity
- Wait list (No Intervention): Wait list

INTERVENTIONS:
Behavioral: Physical activity — 16 weeks
  Arms: Physical activity

SUMMARY:
This randomized controlled trial investigated 12 weeks of physical activity or to 12 weeks in a waiting control condition in youth aged 15 to 24 years old affected by displacement.

DETAILED DESCRIPTION:
In 2020, the Olympic Refuge Foundation (ORF) initiated Game Connect, a sport-for-protection project in Uganda. The current study lasted from September 2022 to August 2023. The project was executed by a consortium led by non-governmental organizations including AVSI Foundation, Right to Play, Youth Sport Uganda, the Uganda Olympic Committee, and the United Nations High Commissioner for Refugees. Included districts were Kampala, Rwamwanja, Palabek, Adjumani, and Kyangwali as they host the largest refugee settlements. Also the surrounding host communities were included. A total of 1,912 potential villages that could be targeted were identified, some of which were grouped in clusters. The decision to cluster villages was influenced by factors such as the limited number of young people in some villages and proximity of households to each other despite living in different villages. In total, 869 villages out of the 1,912 were at random selected for inclusion in the program. Block randomization was applied to ensure equal representation across the targeted districts. Following selection of the villages, all youth in selected villages were identified. Eligible participants in the selected 869 villages of the five catchment areas were: (a) young displaced or host-community adolescents and young adults aged 15 to 24 years, and (b) at least mild symptoms of anxiety and/ or depression, defined as a Patient Health Questionnaire -9, adolescent version (PHQ-9-A) (Spitzer et al., 1999) and / or the Generalized Anxiety Disorder-7 (GAD-7) (Spitzer et al., 2006) score of 5 or higher. Those with severe depression (PHQ-9-A≥20) and / or anxiety (GAD-7≥15) were eligible to participate, but additionally referred to local services for specialized support. Eligible young people were at random allocated to either 12 weeks of physical activity or to 12 weeks in a waiting control condition. All participants completed at baseline and immediately post-intervention the interviewer-administered PHQ-9-A (Spitzer et al., 1999) and GAD-7 (Spitzer et al., 2006). An independent team of well-trained research assistants performed the interviews to minimize potential bias. The research assistants were recruited locally from refugee settlements and surrounding host communities. Data collection tools were pretested to ensure coherence and understandability of questions before the actual data collection commenced. Ethical approval was obtained from the Makerere University School of Social Sciences Research Ethics Committee and the Uganda National Council for Science and Technology. Informed written assent was obtained from all participants. Consent was secured from the current caregivers of youths aged 15-17 years.

ELIGIBILITY:
Inclusion Criteria:

a) young displaced or host-community adolescents and young adults aged 15 to 24 years, and (b) at least mild symptoms of anxiety and/ or depression, defined as a Patient Health Questionnaire -9, adolescent version (PHQ-9-A) (Spitzer et al., 1999) and / or the Generalized Anxiety Disorder-7 (GAD-7) (Spitzer et al., 2006) score of 5 or higher

Exclusion Criteria:

a) young displaced or host-community adolescents and young adults younger than 15 and older than 24 years, and (b) no symptoms of anxiety and/ or depression, defined as a Patient Health Questionnaire -9, adolescent version (PHQ-9-A) (Spitzer et al., 1999) and / or the Generalized Anxiety Disorder-7 (GAD-7) (Spitzer et al., 2006) score lower than 5

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 866 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | 2 weeks
Generalized Anxiety Disorder -7 | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Latimer, Study Director — Olympic Refuge Foundation
Locations (1):
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No